CLINICAL TRIAL: NCT01958944
Title: Phase II Prospective, Open Labeled, Multi-Center, Evaluation of the Safety and Tolerability of Nitric Oxide Given Intermittently Via Inhalation to Subjects With Cystic Fibrosis
Brief Title: Evaluation of the Safety and Tolerability of Inhaled Nitric Oxide to Subjects With Cystic Fibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beyond Air Inc. (Industry)
Collaborators: Soroka University Medical Center (Other); Schneider Children's Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIT_ CP_ CF 01
Record Dates: First submitted 2013-10-06; First posted 2013-10-09 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Cystic Fibrosis
Keywords: CF; Cystic Fibrosis; NO; nitric oxide; inhalation
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Aspiration | interventions — Nitric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nitric oxide + standard treatment (Experimental): Inhalation of 160 ppm NO for 30 minutes, 3 times daily, for a duration of 10 working days with the exclusion of weekend days (Friday & Saturday) in which no treatment under this study will be provided.
  Interventions: Drug: Nitric oxide

INTERVENTIONS:
Drug: Nitric oxide

SUMMARY:
Cystic Fibrosis is defined as a genetic disorder affecting approximately 100,000 individuals worldwide. CF is caused by mutations in the CF Transmembrane Conductance Regulator (CFTR) gene. CF patients are highly prone to environmental opportunistic bacterial infections leading to prolonged and chronic lung infections. This results in reduction in the life expectancy of CF patients due to excessive lung tissue destruction.

Nitric Oxide (NO) is a naturally produced antimicrobial agent which is part of the innate immune defense system of the lung. Both in vitro and in vivo studies had shown clearly that NO acts against a wide variety of microbes including drug resistant bacteria as well as viruses and fungi. Building on a successful phase I safety trial, the team aims to develop a combined drug-device strategy to combat lung infections caused by biofilm-forming bacteria. Unlike other inhaled drugs, NO is also a smooth muscle relaxant and avoids the concomitant bronchial constriction often associated with inhaled antibiotics. An added benefit of NO therapy is its mucolytic activity. We suggest that the combine broad spectrum antimicrobial activity, signaling and mucolytic properties of NO, delivered to the lungs of CF patients, will be directed at reducing bacterial resistance, microbial burden and biofilms as well as resulting in improved airway clearance of viscid sputum.

Primary Objectives: Assess the safety and the tolerability of NO intermittent inhalation treatment in ≥10 years old CF subjects. Secondary Objective: Assess the improvement in forced expiratory volume in 1 second (FEV1) before and after NO intermittent inhalation. Up to 10 subjects with Cystic Fibrosis will be enrolled into the study.

Treatment administration: The subjects will receive intermittent inhalation of NO in addition to standard treatment for 10 working days (no NO treatment will be given to the subjects during weekend days). The subjects will be asked to attend the CF clinic once a week for a period of two weeks in order to evaluate the parameters related to the study. Oxygen (O2), NO, nitrogen dioxide (NO2) and fraction of inspired oxygen (FiO2) delivered to the patient will be continuously monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects (Male or female) ≥10 years old
2. Confirmed diagnosis of CF
3. Resting awake oxygen saturation of at least 92% in room air
4. Approved and signed informed consent:

   1. Subject aged over 10 years old (10 included) -

      * signed an informed consent by the subject
      * Parents/ legal guardian signed informed consent.
   2. Subject aged over 18 years old (18 included) - • signed an informed consent by the subject
5. 80% ≥FEV1≥ 30%
6. Confirmed to be colonized with Pseudomonas aeruginosa

Exclusion Criteria:

1. Subjects younger than 10 years old
2. FEV1< 30% or FEV1> 80%
3. Pulmonary exacerbation resulting in antibiotic treatment (except prophylactic antibiotics) within1 month before enrollment
4. Subject is pregnant (when applicable, a negative pregnancy test result must be verified prior to enrollment and during treatment)
5. Subjects diagnosed with methemoglobinemia, immunodeficiency and/ or heart disease.
6. Use of an investigational drug within 30 days prior enrolment and/ or the subject is expected to participate in a new study within three months from enrollment to this study.
7. History of frequent epistaxis (>1 episode/month)
8. Significant hemoptysis within 30 days (≥ 5 mL of blood in one coughing episode or > 30 mL of blood in a 24 hour period)
9. Methemoglobin level>3% at screening
10. Patients on systemic steroids (1mg/kg or > 20mg of prednisone per day) within 30 days of screening;
11. Smokers;
12. History of illicit drug or medication abuse within 1 year of screening ;
13. history of lung transplantation;
14. Patients treated for high blood pressure
15. Subjects cannot comply with the study design
16. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the subject or the quality of the data.
17. The subject is identified by the investigator as being unable or unwilling to perform study procedures.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Met-Hemoglobin percentage (MetHb)associated with inhaled NO | 1 month
Number of participants with adverse events associated with inhaled NO | 1 month
Proportion of subjects (%) who prematurely discontinued the study for any reason | 1 month
Proportion of subjects (%) who prematurely discontinued the study due to adverse events or serious adverse events | 1 month

SECONDARY OUTCOMES:
Comparing the FEV1 improvement of ≥10 years old with CF before and after NO treatment | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Asher Tal, M.D, Principal Investigator — Soroka University Medical Center; Hannah Blau, M.D, Principal Investigator — Schneider Children's Medical Center, Israel
Locations (2):
- Israel (2):
  - Soroka university, Beersheba
  - Schneider Children's Medical Center of Israel, Petach Tikvah